CLINICAL TRIAL: NCT01218997
Title: A Randomized, Open Label, Long-Term, Multi-Center Study of the Safety of Medisorb® Naltrexone
Brief Title: ALK21-006: Long-Term Study of Medisorb® Naltrexone (VIVITROL®)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard L. Silverman, MD / VP, Clinical Development, Alkermes, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK21-006
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Results first posted 2010-12-13 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Alcoholism
Keywords: Alcoholism; Alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medisorb naltrexone 380 mg (VIVITROL) (Experimental)
  Interventions: Drug: Medisorb naltrexone 380 mg
- Oral naltrexone 50 mg (Active Comparator)
  Interventions: Drug: Oral naltrexone 50 mg

INTERVENTIONS:
Drug: Medisorb naltrexone 380 mg — Administered via intramuscular (IM) injection once every 4 weeks for up to 1 year.
  Other Names: VIVITROL® 380 mg; Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 380 mg (VIVITROL)
Drug: Oral naltrexone 50 mg — Tablet taken orally once daily for up to 1 year
  Other Names: Revia®
  Arms: Oral naltrexone 50 mg

SUMMARY:
This was a Phase 3 multicenter randomized, open-label, safety study assessing the safety of repeat doses of Medisorb® naltrexone 380 mg (VIVITROL®) administered for up to 1 year to adults with alcohol and/or opioid dependence as defined by Diagnostic and Statistical Manual of Mental Health Disorders (DSM-IV) criteria. Eligible subjects were randomized in a 6:1 ratio to receive 1 of the following regimens: a single intramuscular (IM) injection of VIVITROL administered once every 4 weeks or oral naltrexone 50 mg administered daily.

DETAILED DESCRIPTION:
Safety evaluations included physical examinations, electrocardiograms (ECGs), laboratory measures (including plasma concentrations of naltrexone and 6β-naltrexol), assessments of injection sites, and adverse events (AEs).

All subjects received psychosocial support at each study visit for the duration of the study, with interim telephone contact 2 weeks after each monthly visit.

ELIGIBILITY:
Primary Inclusion Criteria:

* Current diagnosis of DSM-IV alcohol dependence and/or diagnosis of DSM-IV opiate dependence within 3 months prior to screening
* 18 years or older
* Desire to seek treatment for alcohol and/or opiate abuse/dependence
* Agree to use contraception for the study duration if of childbearing potential
* Written informed consent and willingness to perform study procedures
* Stable address and phone and at least 1 source of contact information (eg, family member, significant other)

Primary Exclusion Criteria:

* Presence of opiates in the urine (as determined by urine drug test) on Day 0 prior to naltrexone treatment
* Clinically significant medical/psychological condition or abnormality at screening (ie, physical examination, electrocardiogram [ECG], hematology or blood chemistry evaluation, or urinalysis findings)
* Clinically significant active hepatitis or hepatic failure evidenced by 1 of the following: aspartate transaminase (AST) or alanine transaminase (ALT) higher than 3 times the upper limit of normal (3xULN), hyperbilirubinemia (bilirubin >10% above ULN), creatine phosphokinase (CPK) higher than 10xULN, prolonged prothrombin time(international normalized ratio ≥1.7), ascites, or esophageal variceal disease
* Manifestation of suicidal ideation, psychotic symptoms (including significant violent behavior), or psychiatric disorders that would compromise ability to complete the study
* Participation in a formal methadone program currently or within prior 3 years
* More than 2 prior medically supervised detoxification treatments in prior 3 years
* Pregnancy or lactation
* Current prescribed opiate therapy, or receipt of opiates within 7 days prior to study drug dosing, or ongoing medical condition likely to require prescribed opiate therapy during study period
* Failed naloxone challenge on Day 0 (the challenge could be repeated up to 2 times, with at least 24 hours between attempts)
* Participation in a clinical trial within 30 days of screening
* Previous enrollment in a VIVITROL clinical trial
* Receipt of any drug product administered as a gluteal injection within 180 days prior to Day 0 or anticipated need for gluteal injections during study period
* Intolerance and/or hypersensitivity to naltrexone, naloxone, or polylactide-co-polymers such as polylactide-co-glycolide (PLG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2003-08; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was monitored to ensure adequate representation of alcohol-dependent and opioid-dependent patients as defined by Diagnostic and Statistical Manual of Mental Health Disorders (DSM-IV) criteria, and was stratified by alcohol dependence alone versus opioid or mixed substance abuse (ie, alcohol and opioid dependence).
Groups:
- Medisorb Naltrexone 380 mg (VIVITROL): Administered once every 4 weeks via intramuscular (IM) injection for up to 1 year.
- Oral Naltrexone 50 mg: Oral tablet taken once each day for up to 1 year.
Period: Overall Study
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone 50 mg
Started | 371 | 65
Completed | 126 | 24
Not Completed | 245 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone 50 mg | Total
Number analyzed (Participants) | 371 | 65 | 436
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 364 | 64 | 428
  >=65 years | 4 | 1 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.2) | 40.5 (11.4) | 40.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 23 | 161
  Male | 233 | 42 | 275
Region of Enrollment [Number; unit: participants]
  United States | 371 | 65 | 436

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-emergent Adverse Event (TEAE) While on Study
Description: A TEAE was defined as any adverse event (AE) that started or worsened on or after the administration of the first dose of study medication through 30 days after the end of study treatment.
Time Frame: up to 1 year
Population: All subjects who received at least 1 dose of study drug are included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone 50 mg
Number analyzed (Participants) | 371 | 65
Participants | 336 | 53

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone 50 mg
Serious Adverse Events (participants affected / at risk) | 49/371 | 5/65
Other Adverse Events (participants affected / at risk) | 336/371 | 53/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380 mg (VIVITROL) (N=371) | Oral Naltrexone 50 mg (N=65)
Alcoholism (Psychiatric disorders) | 10 | 3
Drug dependence (Psychiatric disorders) | 3 | 1
Suicidal ideation (Psychiatric disorders) | 4 | 0
Suicide attempt (Psychiatric disorders) | 4 | 0
Depression (Psychiatric disorders) | 1 | 2
Mood disorder NOS (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Overdose NOS (Injury, poisoning and procedural complications) | 2 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture NOS (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Non-accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastro-oesophageal reflux (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Convulsions NOS (Nervous system disorders) | 1 | 0
Ischaemic stroke NOS (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Injection site necrosis (General disorders) | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar disc lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical adenitis (Blood and lymphatic system disorders) | 1 | 0
Gastroenteritis NOS (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion spontaneous NOS (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Drug abuser NOS (Social circumstances) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Hypertension NOS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380 mg (VIVITROL) (N=371) | Oral Naltrexone 50 mg (N=65)
Nausea (Gastrointestinal disorders) | 75 | 19
Vomiting NOS (Gastrointestinal disorders) | 32 | 7
Diarrhoea NOS (Gastrointestinal disorders) | 18 | 6
Abdominal pain NOS (Gastrointestinal disorders) | 19 | 3
Dyspepsia (Gastrointestinal disorders) | 10 | 5
Nasopharyngitis (Infections and infestations) | 40 | 11
Upper respiratory tract infection NOS (Infections and infestations) | 40 | 5
Influenza (Infections and infestations) | 22 | 7
Sinusitis NOS (Infections and infestations) | 24 | 3
Urinary tract infection NOS (Infections and infestations) | 23 | 3
Insomnia (Psychiatric disorders) | 41 | 7
Depression (Psychiatric disorders) | 36 | 8
Anxiety NEC (Psychiatric disorders) | 29 | 6
Alcoholism (Psychiatric disorders) | 11 | 4
Headache NOS (Nervous system disorders) | 58 | 11
Dizziness (Nervous system disorders) | 31 | 11
Fatigue (General disorders) | 33 | 11
Injection site pain (General disorders) | 32 | 0
Influenza like illness (General disorders) | 20 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 2
Blood creatinine phosphokinase increased (Investigations) | 20 | 2
Laceration (Injury, poisoning and procedural complications) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should a PI wish to disclose results, the Sponsor will review the results communications prior to public release and can embargo results communications for a period of at least 30 days prior to the submission, for review and approval. Revisions will be negotiated in good faith by the Investigator and Sponsor and may be submitted for publication or disclosed by the Investigator only following receipt of written approval from the Sponsor.